CLINICAL TRIAL: NCT02135484
Title: An Observation, Open Label Study of Alpharadin (Radium 223) in Patients With Castrate Resistant Prostate Cancer Bone Metastases
Brief Title: Radium 223 in Castrate Resistant Prostate Cancer Bone Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry); Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0933; NCI-2014-02016 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Results first posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Adenocarcinoma of the prostate; Castrate resistant prostate cancer; CRPC; Skeletal metastases; Alpharadin; Xofigo; Radium-223 chloride; Radium-223 dichloride
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alpharadin (Experimental): Participants treated with standard dosing of Alpharadin 50 kBq (0.0014 mCi)/kg body weight, administered by slow intravenous injection over 1 minute every 4 weeks for 6 cycles (6 doses total).
  Interventions: Drug: Alpharadin

INTERVENTIONS:
Drug: Alpharadin — 50 kBq (0.0014 mCi)/kg body weight, administered by slow intravenous injection over 1 minute every 4 weeks for 6 cycles (6 doses total).
  Other Names: Xofigo; Radium-223 chloride; Radium-223 dichloride

SUMMARY:
The goal of this clinical research study is to learn more about how the study drug alpharadin (Radium-223) works in patients who have CPRC that has spread to the bone.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive radium-223 by vein over about 1 minute at the beginning of every study cycle for 6 cycles. Every 4 weeks is a study cycle.

You will need to be well hydrated before each dose by drinking at least 2-3 cups (8 ounces each) of water.

Do not take additional drugs, including over-the-counter products and herbal/alternative drugs, during the study without talking with the study doctor first.

Study Visits:

You will have a study visit before each dose of radium-223. The following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 3-4 tablespoons) will be drawn for routine and biomarker tests, as well as to check your PSA and testosterone levels.
* Urine will be collected for biomarker testing.

At Week 12, you will have bone marrow biopsy and aspiration performed to check the status of the disease and for biomarker testing.

At Week 24 the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 3-4 tablespoons) will be drawn for routine tests, as well as to check your PSA and testosterone levels.

Length of Study:

You may receive the study drug for up to 6 doses. You will be taken off study early if the disease gets worse, if you have intolerable side effects, if your study doctor thinks it is in your best interest to stop, or if you are unable to follow study directions.

End of Treatment Visit:

After you stop receiving the study drug for any reason, the following tests and procedures will be performed:

* You will have a physical exam.
* You will have a sodium fluoride PET/CT scan to check the status of the disease.
* Blood (about 3-4 tablespoons) will be drawn for routine and biomarker tests, as well as to check your PSA and testosterone levels.
* Urine will be collected for biomarker testing.
* You will have a bone marrow aspiration and biopsy performed for biomarker testing.

Long-Term Follow-Up:

The study staff will check up on you about every 6 months after your last dose of study drug. This will consist of a phone call, an e-mail, or a review of your medical records. If you are contacted by phone, the call will last about 5 minutes.

This is an investigational study. Radium-223 is FDA approved and commercially available for the treatment of metastatic CRPC that has spread to the bones but not to other organs. It is investigational to look for biomarkers that may be related to CRPC in patients who are receiving radium-223.

The study doctor can explain how the study drug is designed to work.

Up to 25 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven adenocarcinoma of the prostate with evidence for skeletal metastases on bone scan and/or CT scan and symptoms judged to be related to bone metastases
2. Eastern Cooperative Oncology Group (ECOG) performance status < 2. (Karnofsky Performance Status >/= 50%)
3. Serum testosterone levels < 50ng/ml
4. Ongoing gonadal androgen deprivation therapy with Luteinizing Hormone-Releasing Hormone (LHRH) analogues or orchiectomy. Patients, who have not had an orchiectomy, must be maintained on standard dosing of LHRH analogue therapy at appropriate frequency for the duration of the study
5. Life expectancy of at least 12 weeks (3 months)
6. Discontinue any steroids prescribed to specifically treat prostate cancer (for e.g as a secondary hormonal manipulation or for cord compression) > 4 weeks prior to study drug. Steroids chronically prescribed for a non-cancer-related illness [e.g. asthma or chronic obstructive pulmonary disease (COPD)] that is well controlled with medical management are permissible to an equivalent of <10 mg Prednisone daily. Note: Steroids may be administered during the study as supportive care
7. Laboratory Requirements: a.) white blood cell (WBC) count > 3,000/ul; b.) Absolute Neutrophil Count (ANC) > 1,500/ul; c.) Hemoglobin >/= 8.0 g/dL independent of transfusion; d.) Platelet count >/= 100,000/uL; e.) Serum albumin >/= 3.0 g/dL; f.) Calculated or measured creatinine clearance > 30 mL/min
8. All acute toxic effects of any prior treatment have resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.0 Grade 1 or less at the time of signing the Informed Consent Form (ICF)
9. Patient must be willing and able to comply with protocol requirements. All patients must sign an informed consent indicating that they are aware of the investigational nature of this study
10. Patients must also have signed an authorization for the release of their protected health information

Exclusion Criteria:

1. Treatment with cytotoxic chemotherapy within previous 4 weeks of protocol treatment, or failure to recover from AEs due to cytotoxic chemotherapy administered more than 4 weeks prior to protocol treatment (however, ongoing neuropathy is permitted)
2. Received systemic therapy with radionuclides (e.g., strontium-89, samarium-153, rhenium-186, or rhenium-188, or Ra-223 dichloride) for the treatment of bony metastases
3. Other malignancy treated within the last 3 years (except non melanoma skin cancer or low-grade superficial bladder cancer)
4. Visceral metastases as assessed by abdominal or pelvic computed tomography (CT) (or other imaging modality)
5. Known brain metastases
6. Lymphadenopathy exceeding 6 cm in short-axis diameter
7. Any size pelvic lymphadenopathy if it is thought to be a contributor to concurrent hydronephrosis
8. Imminent spinal cord compression based on clinical findings and/or magnetic resonance imaging (MRI). Treatment should be completed for spinal cord compression
9. Any other serious illness or medical condition, such as but not limited to: a) Any infection >/= National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0 Grade 2; b) Cardiac failure New York Heart Association (NYHA) III or IV; c) Crohn's disease or ulcerative colitis; d) Bone marrow dysplasia; e) Fecal incontinence
10. Inability to comply with the protocol and/or not willing or not available for follow-up assessments
11. Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation
12. Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization) other than Ra 223 dichloride
13. Prior use of Ra-223 dichloride, Strontium or Samarium
14. Concurrent use of another investigational drug or device therapy (i.e., outside of study treatment) during, or within 4 weeks of trial entry (signing of the informed consent form)
15. Major surgery within 30 days prior to start of study drug

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-09-19 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Araujo, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Corn PG, Yu G, Fan Y, Zhang M, Troncoso P, Surasi DS, Liu S, Ajani JA, Logothetis CJ, Wang G, Panaretakis T, Lin SH. Spatial immune profiling of bone-metastatic castration-resistant prostate cancer reveals radium-223 immunomodulates the bone-tumor microenvironment. Prostate Cancer Prostatic Dis. 2025 Dec 26. doi: 10.1038/s41391-025-01069-1. Online ahead of print. PMID 41454189
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 27 participants consented, 2 participants ineligible (1) withdrawal by subject and (1)screen failure.
Period: Overall Study
Arm/Group | Alpharadin
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alpharadin
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 66 [46 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 25
Prostate Specific Antigen (PSA) Levels [Median (Full Range); unit: ng/mL] — PSA is produce by normal and cancerous prostate tissue. PSA levels are often elevated in men with prostate cancer.
  ng/mL | 26.9 [0.1 to 4170]
Total Alkaline Phosphatase Level [Median (Full Range); unit: U/L] — Elevated total alkaline phosphatase is an indication that the prostate cancer has spread to bones. Normal range 38 126 U/L
  U/L | 489 [64 to 681]
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG measure a participant's daily living abilities. All participants in this trial are grade 0 and grade 1 Grade 0: Fully active Grade 1: light house work and office work. Restricted in physically strenuous activity
  Participants
    Grade 0 | 12
    Grade 1 | 13
Gleason Score [Count of Participants; unit: Participants] — Gleason score grades prostate cancer based on the severity of the cancer The scores range from 2 -10. The higher the score the more severe the cancer. Gleason Score of 6 is the lowest cancer grade. Gleason score of 7 is an intermediate grade Gleason score of 8 -10 is a high grade
  Participants
    Score of 7 | 3
    Score of 8 | 5
    Score of 9 | 14
    Score of 10 | 1
    Unknown | 2
Extent of Bone Metastases [Count of Participants; unit: Participants] — Participants are put into two categories.Those with less that 20 bone metastases. Those with more than 20 bone metastases.
  Participants
    Less than 20 | 8
    More than 20 | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (Favorable and Unfavorable )
Description: Overall survival is measured in months from the time of enrollment until death. Participants who survived longer then the median survival rate of 24.3 months were assigned favorable survival. Participants who survived less than 24.3 months were assigned unfavorable survival.
Time Frame: 3.6 years
Measure: Median (Full Range); unit: months
Arm/Group | Alpharadin
Number analyzed (Participants) | 25
months
  Unfavorable Survival | 13.9 [3.3 to 23.1]
  Favorable Survival | 36.3 [24.3 to 43.1]

ADVERSE EVENTS:
Time Frame: adverse event data collected up to 3 years
Arm/Group | Alpharadin
All-Cause Mortality (participants affected / at risk) | 19/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 13/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpharadin (N=25)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Fatigue (General disorders) | 8 (8)
Platelet count decreased (Investigations) | 3 (3)
White blood cell decreased (Investigations) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT02135484/Prot_SAP_000.pdf